CLINICAL TRIAL: NCT06712641
Title: Aminoglycosides in Early Sepsis (AGES): A Randomized Pragmatic Clinical Trial Comparing Gentamicin and Narrow Spectrum Betalactams to Broad Spectrum Betalactams as Empirical Treatment in Patients With Suspected Sepsis
Brief Title: Aminoglycosides in Early Sepsis
Acronym: AGES
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Ullevaal University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Nakrem Lyngbakken, Postdoctoral fellow, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-519797-39-00
Record Dates: First submitted 2024-11-27; First posted 2024-12-02 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Sepsis
Keywords: sepsis; antibiotics; aminoglycosides; cephalosporins
MeSH Terms: conditions — Sepsis | interventions — Gentamicins; Cefotaxime; Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gentamicin + narrow spectrum betalactam (Active Comparator): Empirical therapy for suspected community-acquired sepsis with gentamicin + narrow spectrum betalactam (either one of penicillin, ampicillin, or cloxacillin)
  Interventions: Drug: Gentamicin + narrow spectrum betalactam
- Cefotaxime or piperacillin-tazobactam (Active Comparator): Empirical therapy for suspected community-acquired sepsis with broad spectrum betalactam (either one of cefotaxime or piperacillin-tazobactam)
  Interventions: Drug: Cefotaxime; Drug: Piperacillin-tazobactam

INTERVENTIONS:
Drug: Gentamicin + narrow spectrum betalactam — Empirical therapy for suspected community-acquired sepsis with gentamicin + narrow spectrum betalactam (either one of penicillin, ampicillin, or cloxacillin)
  Arms: Gentamicin + narrow spectrum betalactam
Drug: Cefotaxime — Empirical therapy for suspected community-acquired sepsis with cefotaxime
  Arms: Cefotaxime or piperacillin-tazobactam
Drug: Piperacillin-tazobactam — Empirical therapy for suspected community-acquired sepsis with piperacillin-tazobactam
  Arms: Cefotaxime or piperacillin-tazobactam

SUMMARY:
Norwegian guidelines for empirical antibiotic therapy in suspected community acquired sepsis recommend the combination of narrow spectrum betalactam and aminoglycoside as the first choice, but broad spectrum betalactams are considered equally appropriate, effective, and safe. However, fear of renal complications due to gentamicin and concern for lacking evidence for efficiency commonly leads to the use of broad spectrum betalactam therapy, a larger driver of antibiotic resistance.

In patients with suspected community acquired sepsis, the investigators hypothesize that empirical combination therapy with narrow spectrum betalactams and aminoglycosides is safe and non-inferior to empirical therapy with broad spectrum betalactams. More specifically, the investigators hypothesize that the proportion of patients with acute kidney injury or death will be similar between these two treatment groups. Furthermore, the investigators hypothesize that the aminoglycoside-based regimen has lesser impact on the gut microbiome. Antimicrobial resistance is one of the most urgent health threats of our time, and Norwegian hospitals were required but failed to reduce the use of broad-spectrum antibiotics with 30% by the end of 2020. In this context, novel initiatives aiming at reducing use of antibiotics are direly needed.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized
* Adults 18 year or older
* Clinical suspicion of community acquired sepsis with indication for empirical antibiotic therapy
* National Early Warning Score 2 (NEWS2) ≥ 5
* Signed informed consent must be obtained and documented according to ICH GCP, and national/local regulations

Exclusion Criteria:

* Established chronic kidney failure (eGFR < 30 ml/min/1.73m2)
* Presentation with septic shock with multiorgan failure
* Suspicion of condition necessitating specific antimicrobial therapy (e.g. atypical pneumonia, fungal infection, parasitic infection, mycobacterial infection)
* Current or recent use of nephrotoxic drugs (e.g cisplatin within previous 2 months)
* Suspected or confirmed carrier of extended spectrum betalactamase (ESBL) producing bacteria, methicillin-resistant Staphylococcus aureus (MRSA), or other drug-resistant microbes necessitating specific antimicrobial therapy
* Multiple myeloma
* Renal transplantation
* Renal replacement therapy
* Myasthenia gravis
* Known hypersensitivity to any of the study drugs
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1900 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | Up to 30 days after randomization
  All-cause mortality up to 30 days after randomization
30-day acute kidney injury | Up to 30 days after randomization
  Any acute kidney injury up to 30 days after randomization

SECONDARY OUTCOMES:
In-hospital mortality | During index hospitalization (commonly up to 30 days)
  All-cause mortality during index hospitalization
Duration of hospital stay | During index hospitalization (commonly up to 30 days)
  Duration of index hospitalization (days)
Duration of intensive care stay | During index hospitalization (commonly up to 30 days)
  Duration of stay in intensive care unit (days)
Duration of ventilator therapy | During index hospitalization (commonly up to 30 days)
  Duration of therapy with invasive mechanical ventilation (days)
Duration of vasopressor therapy | During index hospitalization (commonly up to 30 days)
  Duration of therapy with vasoactive (vasopressor) (days)
Hospital readmissions | Up to 30 days after discharge from index hospitalization
  Readmission after discharge from index hospitalization
Post-discharge mortality | Up to 30 days after discharge from index hospitalization
  All-cause mortality after discharge from index hospitalization
Duration of antibiotic treatment | During index hospitalization (commonly up to 30 days)
  Duration of antibiotic therapy during index hospitalization (days of therapy, DOT)
Gut microbiome composition | During index hospitalization (commonly up to 30 days)
  Impact on the gut microbiome

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital Ullevål, Oslo

IPD SHARING:
Plan to Share IPD: No
The dataset used in this study is not publicly available, as the Data Protection Authority approval and patient consent do not allow for such publication. The study group welcomes initiatives for cooperation and data access may be granted upon application.